CLINICAL TRIAL: NCT06341166
Title: Multiparametric SCores for Prediction of Myocardial fIbrosis in Patients With MITral vAlve pRolapse: the SCIMITAR Trial
Brief Title: Multiparametric SCores for Prediction of Myocardial fIbrosis in Patients With MITral vAlve pRolapse
Acronym: SCIMITAR
Status: Recruiting | Type: Observational
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Humanitas Hospital, Italy (Other); IRCCS Ospedale San Raffaele (Other); Azienda Ulss 2 Marca Trevigiana (Other)
Responsible Party: Sponsor
Other Study IDs: CCM1959
Record Dates: First submitted 2024-03-14; First posted 2024-04-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Mitral Valve Prolapse
MeSH Terms: conditions — Mitral Valve Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Cohort: Prospectively enrolled patients will undergo a complete assessment, as clinically indicated, including clinical evaluation, TTE, rest ECG, 24h ECG-monitoring, and CMR. CMR will be performed no more than 6 months apart from other examinations (TTE, rest ECG, 24h ECG-monitoring).
- Retrospective Cohort: Patients will be enrolled retrospectively, in case they have already performed all examinations between 2016 and 2023

SUMMARY:
This is a multicenter, observational prospective and retrospective study which aims are: 1) to compute a scoring model potentially predictive for the diagnosis of fibrosis by CMR in patients with MVP; 2) to identify specific features that may predispose to ≥ mild VAs or SCD in patients with MVP.

DETAILED DESCRIPTION:
Patients with mitral valve prolapse and non-significant mitral regurgitation generally have a good prognosis. A minority of patients with MVP suffers from ventricular arrhythmias. Different demographic, clinical, and electrocardiographic characteristics, as well as morphological and structural features of the MV were described as potential risk factors for ventricular arrhythmias, among which fibrosis of the left ventricular inferolateral wall and posterior papillary muscle as detected by cardiac magnetic resonance.

As cardiac magnetic resonance has some limitations, it is unknown if and which patients with mitral valve prolapse should undergo cardiac magnetic resonance in routine clinical practice, to search for late gadolinium enhancement as a surrogate for myocardial fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* Echocardiographic diagnosis of mitral valve prolaspe, defined as a systolic displacement of one or both mitral leaflets ≥ 2 mm above the plane of the mitral valve annulus in long-axis views

Exclusion Criteria:

* age< 18 years
* coexistence of other cardiomyopathies or other ≥ moderate valve diseases
* scarce acoustic transthoracic echocardiographic window
* usual contraindications for cardiac magnetic resonance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of mitral valve prolapse by transthoracic echocardiography, independent of mitral regurgitation grade, either affected by Barlow's disease, fibroelastic deficiency, forme frustae of mitral valve prolapse.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2026-06-19 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
Prediction of fibrosis by CMR | June 2026
  Clinical, echocardiographic, electrocardiographic, and 24h-ECG monitoring variables will be collected in order to identify potential predictors of fibrosis as detected by cardiac magnetic resonance (CMR).
  Specifically, the following parameters will be collected.
  * Clinical data:
  * Transthoracic echocardiography parameters:
  * Rest ECG parameters:
  * 24h electrocardiographic monitoring parameters:
  * Ventricular arrhythmias (VAs) will be classified as suggested in the recently published EHRA consensus statement
  * CMR parameters, applying the protocol of the Society of Cardiovascular Magnetic Resonance

SECONDARY OUTCOMES:
Prediction of ≥ mild Ventricular Arrhythmias and/or Sudden cardiac death in mitral valve | June 2026
  Clinical, echocardiographic, electrocardiographic, and CMR variables will be collected in order to identify potential predictors of ≥mild VAs, as defined by the recently published EHRA consensus document.
  An accurate description of these variables and the Units of Measure are the same as those reported in the section "Primary Outcome Measures".
Clinical data | June 2026
  * gender (female/male), and age in years;
  * family history for sudden cardiac death;
  * previous documentation of supraventricular and/or ventricular arrhythmias (VAs);
  * previous secondary prevention ICD implantation, previous transcatheter ablation of VAs;
  * symptoms (history of unexplained syncope/pre-syncope, palpitations, dyspnea, chest pain);
  * signs (mid-systolic click, murmurs of mitral regurgitation);
  * use of anti-arrhythmic drugs and/or beta-blockers.
Transthoracic echocardiography parameters: | June 2026
  * left atrial biplane volume in mL/m2;
  * presence, localization, and end-systolic measurement in millimeters of mitral annular disjunction (MAD);
  * mitral leaflet thickness in millimeters, presence of bileaflet prolapse;
  * mitral regurgitation (MR) grade, quantified by integrating qualitative and quantitative criteria according to the European guidelines;
  * left ventricular (LV) diameters in millimeters, volumes in mL/m2, and ejection fraction in %;
  * presence of curling of the posterolateral LV wall;
  * presence of the Pickelhaube sign at tissue Doppler imaging;
  * right ventricular end-diastolic area in cm2/m2, TAPSE in millimeters, and fractional area change in %;
  * systolic pulmonary artery pressure in mmHg, derived from the peak velocity of the tricuspid regurgitation and from the estimated right atrial pressure.
Rest ECG parameters: | June 2026
  * baseline rhythm (sinus rhythm, atrial fibrillation/flutter, junctional rhythm);
  * PQ and QRS intervals in milliseconds;
  * T wave inversion or biphasic T waves in the inferior and lateral leads;
  * QTc interval in milliseconds;
  * occurrence of premature supraventricular complexes;
  * occurrence of premature ventricular complexes (PVCs).
24h electrocardiographic monitoring parameters: | June 2026
  * baseline rhythm (sinus rhythm, atrial fibrillation/flutter, junctional rhythm);
  * frequency (expressed in absolute number and as percentage of total beats number), and repetitiveness of premature supraventricular complexes;
  * occurrence of atrial fibrillation;
  * frequency (expressed in absolute number and as percentage of total beats number), and repetitiveness of PVCs.
  Ventricular arrhythmias (VAs) will be classified as suggested in the recently published EHRA consensus statement:
  * MILD VAs, defined as ≥ 5% total PVC burden or non-sustained (< 30 seconds) ventricular tachycardia (VT) runs with a heart rate < 120 bpm
  * MODERATE VAs, defined as non-sustained (< 30 seconds) VT runs with a heart rate of 120-179 bpm
  * SEVERE VAs, defined as non-sustained (< 30 seconds) VT runs with a heart rate > 180 bpm or sustained (≥ 30 seconds) VT/ventricular fibrillation.
CMR parameters | June 2026
  * MR grade (based on the regurgitant volume and regurgitant fraction);
  * LV mass in g/m2;
  * biventricular volumes in mL/m2, stroke volumes in mL, and ejection fraction in %;
  * presence of curling of the posterolateral LV wall;
  * presence, localization, end-systolic and end-diastolic measurement in millimeters of MAD;
  * presence and distribution of LGE.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Cardiologico Monzino, Milan, Milan, Italy